CLINICAL TRIAL: NCT05248698
Title: Dry Eye Response to Interval Exercise (High Intensity Aerobic Activity) and Mediterranean Diet
Brief Title: Dry Eye Response to Interval Exercise and Mediterranean Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003553
Record Dates: First submitted 2022-02-07; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Dry Eye; Diet Habit; Physical Inactivity
MeSH Terms: conditions — Dry Eye Syndromes; Feeding Behavior; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): 30 older patient who will complain from dry eye will receive 3-time interval exercise per the week, applied for 30 min with high intensity, plus Mediterranean Diet for 6 months
  Interventions: Behavioral: lifestyle change
- group 2 (Active Comparator): 30 older patient who will complain from dry eye will receive 3-time interval exercise per the week, applied for 30 min with high intensity, for 6 months
  Interventions: Other: exercise

INTERVENTIONS:
Behavioral: lifestyle change — 30 older patient who will complain from dry eye will receive 3-time interval exercise per the week, applied for 30 min with high intensity, plus Mediterranean Diet for 6 months
  Arms: group 1
Other: exercise — 30 older patient who will complain from dry eye will receive 3-time interval exercise per the week, applied for 30 min with high intensity, for 6 months
  Arms: group 2

SUMMARY:
in the recent times, dry eye was found to be correlated sedentary life style, obesity, hypertension. So, changing the sedentary lifestyle is recommended

DETAILED DESCRIPTION:
older patient who will complain from dry eye will be collected. it is planned to recruit 60 elderly (with obesity and hypertension) to be distributed into group 1 (this group will receive 3-time interval exercise per the week, applied for 30 min with high intensity, plus Mediterranean Diet) and group 2 (this group will receive only 3-time interval exercise per the week, applied for 30 min with high intensity). Every group will contain 30 elderly

ELIGIBILITY:
Inclusion Criteria:

* elderly patients with dry eye complaints
* the patients will be obese and hypertensives

Exclusion Criteria:

* heart or respiration problems
* other diagnosed eye or systemic diseases

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 60 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Schirmer's test | 6 months
  tear-production speed test

SECONDARY OUTCOMES:
scoring system for dry eye | 6 months
  it is a questionnaire will assess dry-eye severity
Ocular surface disability index | 6 months
  it is a questionnaire will assess complaints of patients due to severity of dry-eye
tear film break up time testing | 6 months
  it is a test that will assess tear film stabilization
Oxford grading system | 6 months
  a test will examine ocular epithelial damage
blood systole | 6 months
  it will be measured by sphygmomanometer
blood diastole | 6 months
  it will be measured by sphygmomanometer
weight | 6 months
  it will be expressed in kilograms
body mass index | 6 months
  it will be gained by dividing weight of subject on his or her squared height
waist circumference | 6 months
  it will be evaluated by tape measurements of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt